CLINICAL TRIAL: NCT01805063
Title: Effect of Fire Suppression and Emergency Duties on Vascular Function in Firefighters
Brief Title: Effect of Fire Suppression and Emergency Duties on Vascular Function
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 11-SS-0049; PG/11/27/28842 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2013-03-04; First posted 2013-03-05 (Estimated); Last update posted 2024-05-01 (Actual); Status verified 2013-03

CONDITIONS: Vascular Function; Atherothrombosis
Keywords: firefighters; myocardial infarction; endothelial function; thrombosis; fire suppression; non-fire emergency duty; sedentary shift
MeSH Terms: conditions — Thrombosis; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and urine samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Fire suppression: Firefighters will attend for vascular assessments following a night shift where they have performed fire suppression
  Interventions: Procedure: Forearm Vascular Study; Procedure: Badimon Chamber
- Non-fire emergency duty: Firefighters will attend for vascular assessments following a night shift where they have had an emergency response without fire suppression eg. road traffic collision.
  Interventions: Procedure: Forearm Vascular Study; Procedure: Badimon Chamber
- Sedentary shift: Firefighters will attend for vascular assessments following a night shift where they have remained sedentary throughout the shift.
  Interventions: Procedure: Forearm Vascular Study; Procedure: Badimon Chamber

INTERVENTIONS:
Procedure: Forearm Vascular Study — Forearm venous occlusion plethysmography to measure forearm blood flow during intra-arterial infusion of the vasodilators Verapamil (10-100 µg/min), bradykinin (100-1000 pmol/min), sodium nitroprusside (2-8 µg/min) and Acetylcholine (5-20 µg/min).
  Other Names: BK; SNP; ACh; VP
Procedure: Badimon Chamber — Ex-vivo assessment of thrombus formation using the Badimon Chamber

SUMMARY:
Firefighters are at increased risk of death from heart attacks when compared to other emergencyy service professionals whose jobs involve similar components such as emergency call-outs and shift work. In the largest analysis of cause of death amongst on-duty firefighters, firefighter deaths were classified according to the duty performed during the onset of symptoms or immediately prior to any sudden death. The majority of deaths due to a cardiovascular cause (i.e. heart attack) occurred during fire suppression whilst this activity represented a relatively small amount of a firefighters professional time. There was also a risk of death associated with other duties such as emergency non-fire response and physical exertion.

The investigators hypothesize that participation in active fire-fighting duties impairs blood vessel function and increases blood clot formation when compared with non-fire-fighting activities. In this study, healthy career firefighters will be assessed after three periods of duty: fire-suppression, emergency response without fire suppression and following a sedentary shift. The investigators will take blood samples to measure platelet activity (platelets are the particles in blood that help blood clot) and will examine how blood clots outside of the body. The investigators will then perform studies placing small needles in the arm to assess blood vessel function following these duties. By undertaking this comprehensive assessment of blood, blood vessel and heart function the investigators hope to understand the mechanisms whereby the risk of a heart attack, fatal or otherwise, is posed throughout these distinct duties that firefighters undertake on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking healthy firefighters

Exclusion Criteria:

* Current smoker
* History of lung or ischaemic heart disease
* Malignant arrhythmia
* Systolic blood pressure >190mmHg or <100mmHg
* Renal or hepatic dysfunction
* Previous history of blood dyscrasia
* Unable to tolerate the supine position
* Blood donation within the last 3 months
* Recent respiratory tract infection within the past 4 weeks
* Routine medication including aspirin and NSAIDs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be healthy, non-smoking, whole-time firefighters working within Lothian and Borders Fire and Rescue Service
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-01-09 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow measured by venous occlusion plethysmography in response to infused vasodilators | up to 12 hours after exposure

SECONDARY OUTCOMES:
Ex-vivo thrombus formation using the Badimon chamber | up to 12 hours after exposure
Plasma t-PA and PAI concentrations following infusion of bradykinin | During forearm study, up to 12 hours after exposure

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, MD PhD, Study Chair — University of Edinburgh; Nicholas L Mills, MBChB PhD, Study Director — University of Edinburgh; Amanda L Hunter, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh Clinical Research Facility, Edinburgh, United Kingdom